CLINICAL TRIAL: NCT02511938
Title: Introducing Child Menus in Restaurants to Improve Access to Healthier Foods
Brief Title: Kids' Choice Restaurant Program
Acronym: KCRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Guadalupe X. Ayala, Associate Dean, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R21HD071324 (NIH)
Record Dates: First submitted 2015-07-21; First posted 2015-07-30 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Childhood Obesity
Keywords: childhood obesity; restaurant; away from home foods
MeSH Terms: conditions — Pediatric Obesity | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Menu Only intervention (Experimental): Restaurants will receive a new healthy kids' menu
  Interventions: Other: Menu Only
- Menu Plus Intervention (Experimental): Restaurants will receive a new healthy kids' menu, supporting marketing materials, and brief trainings for customer service staff and kitchen staff to support and promote the new menu items.
  Interventions: Other: Menu Plus intervention

INTERVENTIONS:
Other: Menu Only — Restaurants will collaborate with project to develop and introduce new healthy kid's menu items. Project will provide recipes, preparation support, nutritional information, and printed menus to restaurants.
  Arms: Menu Only intervention
Other: Menu Plus intervention — Restaurants will collaborate with project to develop and introduce new healthy kid's menu items. Project will provide recipes, preparation support, nutritional information, and printed menus to restaurants. In addition, project will provide promotional materials and brief restaurant staff trainings to promote the new menu.
  Arms: Menu Plus Intervention

SUMMARY:
This study will introduce healthy child menu items into 8 independent full service restaurants in San Diego County. The restaurants will be assigned either to receive new, healthy kids' menu items or to receive the new menu items in addition to marketing materials and staff trainings to support promotion of these new menu items. The primary outcome for the study is sales of kids' menu items. Additional customer observation and interview data will be collected, as well as manager interviews and restaurant environment assessments. Process evaluation measures will also evaluate the implementation of the intervention.

DETAILED DESCRIPTION:
The purpose of the study is to assess the efficacy of an intervention to improve access to healthier foods by introducing or changing child menus in restaurants. We propose recruiting 8 independent full service restaurants, either with or without existing child menus. Recruitment will occur in waves of two restaurants per wave for a total of four waves. Restaurants will be matched on key criteria such as whether they have a child menu and restaurant size based on seating (categorized as small -to- medium or large). Matched restaurants will be randomized to either an 8--week menu--only intervention or a menu--plus intervention that will occur at the same time. The menu--only intervention will involve working with the restaurant to add new healthy child menu items to their menus. The menu--plus intervention will involve working with the restaurants to add new healthy child menu items tailored to their menus, along with promotional materials and restaurant employee trainings to encourage customers to select these menu items. Weekly detailed sales data (reported by menu item) at baseline for one month, ongoing in all restaurants during 8-week intervention, and for one month at post intervention for all restaurants will be gathered and serve as the primary outcome of interest. Additionally, biweekly observations and customer interviews in each restaurant during one month pre--intervention phase, over 8--week intervention period, and during one month post-intervention phase to capture how orders are placed and what is ordered and reported to be consumed by the child. We will also assess the feasibility and fidelity of the intervention using manager interview data (baseline and post--intervention), restaurants audits (baseline, once during the intervention, and at post--intervention), and process evaluation measures (weekly during 8-week intervention). The study is not designed to provide a direct benefit to the participants and no such benefits can be guaranteed; however, participants may learn more about current public health research and efforts to understand child ordering and consumption behaviors in restaurants. This study may benefit independent restaurants as the findings will contribute to designing evidence--based approaches to improving the nutritional quality of child menu offerings and will help researchers to understand ordering and consumption behaviors for children in restaurants. This study presents minimal risks to the participants.

ELIGIBILITY:
For customer observations and interviews:

Inclusion Criteria:

* Restaurant dining parties having at least one adult 18 or older and one child in party who appears to be between the ages of 3--17 years
* Dining parties including no more than six people
* Party speaks English and/or Spanish

Exclusion Criteria:

* Party does not speak English and/or Spanish
* Parties larger than six people

For restaurant manager interviews:

Inclusion Criteria:

* At least 18 years of age
* Has worked at restaurant at least 4 months
* Works at least 20 hours per week for the restaurant
* Plans to continue working at the restaurant for at least 6 months
* Speaks and writes English and/or Spanish

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2013-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Sales ($) of kids' menu items | weekly throughout study period (4 wk baseline, 8 wk Ix phase, 4 week post-ix)
  Change in weekly sales ($) of kids' menu items as a proportion of total restaurant sales between baseline, intervention period, and post-intervention

SECONDARY OUTCOMES:
Customer observations/interviews | every other week throughout study period (4 wk baseline, 8 wk Ix phase, 4 week post-ix)
  change in child customer ordering behavior, decision making, and consumption between baseline, intervention period, and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe X Ayala, PhD, MPH, Principal Investigator — San Diego State University
Locations (1):
- SDSU Research Foundation, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ayala GX, Castro IA, Pickrel JL, Williams CB, Lin SF, Madanat H, Jun HJ, Zive M. A restaurant-based intervention to promote sales of healthy children's menu items: the Kids' Choice Restaurant Program cluster randomized trial. BMC Public Health. 2016 Mar 10;16:250. doi: 10.1186/s12889-016-2892-5. PMID 26965639